CLINICAL TRIAL: NCT00491894
Title: A Six-Month, Multi-Center, Open-Label Study to Assess the Safety and Efficacy of Oral Glycopyrrolate Liquid for the Treatment of Pathologic (Chronic Moderate to Severe) Drooling in Pediatric Patients 3 to 18 Years of Age With Cerebral Palsy or Other Neurologic Conditions
Brief Title: Safety and Efficacy Study of Oral Glycopyrrolate Liquid for the Treatment of Pathologic (Chronic Moderate to Severe) Drooling in Pediatric Patients 3 to 18 Years of Age With Cerebral Palsy or Other Neurologic Conditions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Shionogi Clinical Trials Administrator, Shionogi
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sc-GLYCO-06-01; NCT00425087 (obsolete NCT alias)
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-04

CONDITIONS: Cerebral Palsy; Neurological Conditions; Mental Retardation; Sialorrhea
Keywords: Mental Retardation; Neurological Impairment; Cerebral Palsy; Drooling; Neurological Conditions
MeSH Terms: conditions — Cerebral Palsy; Intellectual Disability; Sialorrhea; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Chronic Drooling (Other): Arm receiving study drug
  Interventions: Drug: Oral Glycopyrrolate Liquid

INTERVENTIONS:
Drug: Oral Glycopyrrolate Liquid — Study medication is administered three times a day at 7-8 AM, 1-2 PM, and 7-8 PM by the parent/caregiver

SUMMARY:
This is an open-label clinical research study of an oral glycopyrrolate liquid for the treatment of chronic moderate to severe drooling in patients with cerebral palsy or other neurological conditions. Patients participating in the study will receive oral glycopyrrolate liquid (1 mg/5 ml) three times a day (TID) for study duration of 24 weeks. After a washout, screening, and 2-day baseline period, patients will be enrolled in a 4-week dose titration period. Glycopyrrolate liquid doses will be titrated using dose levels in the Dose Titration Schedule. Titration will begin at 0.02 mg/kg per dose TID and sequentially increased in 0.02 mg/kg per dose increments TID every 5-7 days during the first four weeks until optimal individualized response is obtained for each patient or a maximum dose of 0.1 mg/kg TID is reached, not exceeding 3 mg TID or Dose-level 5 in the Dose Titration Schedule, whichever is lesser. Optimal dose for each patient is the dose at which he/she is receiving the maximum benefit from the study drug (greatest improvement in drooling) while experiencing minimum side effects. All patients will receive close attention by study staff throughout the study.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, patients must meet the following criteria:

* Male or female, weighing at least 13 kilograms (27 pounds), aged 3 through 18 years
* Diagnosis of cerebral palsy and/or mental retardation or any other neurologic impairment or condition (cognitively capable and cognitively impaired patients may be enrolled)
* Chronic drooling in the absence of treatment to the extent that the chin or clothing becomes wet on most days by confirming the Modified Teacher's Drooling Scale score ≥ 5
* Must be living in a situation where reliable parents/caregivers are willing and capable of administering medications, as determined by the investigator
* Written informed consent signed by the parent or legally acceptable representative
* Written assent signed by the age-appropriate patient if mentally capable, as determined by the investigator, and required by the site's Institutional Review Board
* If female of childbearing potential, the patient must have a negative pregnancy test at screening and Visit 2
* If female of childbearing potential and sexually active, she must use a medically acceptable form of contraception

Exclusion Criteria:

Patients are excluded from this study if they meet any of the following criteria:

* Patients who used glycopyrrolate within approximately 24 hours prior to the start of the baseline period, which began on Day -2
* Patients who used prohibited medications within 5 plasma half-lives of the medication prior to the start of the baseline period
* Patients injected with intrasalivary gland botulinum toxin within 10 months prior to the start of the baseline period
* Patients using intraoral devices or prosthetics for the treatment of drooling within 1 week prior to the start of the baseline period
* Patients receiving acupuncture for the treatment of drooling or who have received acupuncture for the treatment of drooling within 3 months prior to the start of the baseline period
* Patients who have medical conditions contraindicating anticholinergic therapy including gastrointestinal reflux, narrow-angle glaucoma, obstructive uropathy, obstructive disease of the gastrointestinal tract (i.e., delayed gastric emptying, pyloroduodenal stenosis, etc.), paralytic ileus, intestinal atony, vesicoureteral reflux, reactive airway disease, myasthenia gravis, hyperthyroidism, cardiac arrhythmias and/or tachycardia, and/or clinically significant electrocardiogram abnormalities, as determined by the investigator
* Patients who have a known contraindication to the study medication, including allergy to the study medication or any of its components
* Patients who have poorly controlled seizures defined as daily seizures
* Patients who have a history of obstructive disease of the gastrointestinal tract (i.e., intestinal obstruction)
* Patients who have clinically significant hepatic or renal impairment, at the discretion of the investigator
* Patients who are pregnant or breastfeeding
* Patients who have received any investigational drugs within 30 days of study entry
* Patient, families, or parents/caregivers who are expected to be non-compliant with the study procedures, as judged by the investigator
* Patients who are unable to meet the requirements of the study for any reason, as determined by the investigator
* Patients who have unstable mental disease, as determined by the investigator

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (7):
- United States (7):
  - Rocky Mountain Pediatrics, Lakewood, Colorado
  - Child Neurology Associates, PC, Atlanta, Georgia
  - St. Mary's for Children, Bayside, New York
  - Akron's Childrens, Akron, Ohio
  - Hattie Larltham Center for Children with Disabilities, Mantua, Ohio
  - The Children's Center, Bethany, Oklahoma
  - Alamo City Clinical Research, San Antonio, Texas

REFERENCES:
- [Derived] Zeller RS, Lee HM, Cavanaugh PF, Davidson J. Randomized Phase III evaluation of the efficacy and safety of a novel glycopyrrolate oral solution for the management of chronic severe drooling in children with cerebral palsy or other neurologic conditions. Ther Clin Risk Manag. 2012;8:15-23. doi: 10.2147/TCRM.S26893. Epub 2012 Jan 25. PMID 22298950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on April 03, 2007 and last patient completed on May 30, 2008
Pre-assignment Details: After a washout and screening period, and 2-day baseline period, patients were enrolled in a 4-week dose titration period which commenced with the goal of identifying an optimal 3 times daily maintenance dose for each patient. The resulting individualized optimal maintenance dose was to be administered for the remainder of the 24-week study
Groups:
- Patients With Chronic Drooling: A 4-week dose titration period until an optimal individualized response was obtained for each patient or a maximum dose of 0.1 mg/kg/dose was reached. Doses were not to exceed 3.0 mg/kg TID
Period: Overall Study
Arm/Group | Patients With Chronic Drooling
Started | 137
Completed | 103
Not Completed | 34
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 5
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 2
Not completed — Other-Failed to meet any criteria | 2
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 2
Not completed — Other-Intake of prohibited medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Chronic Drooling
Number analyzed (Participants) | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 137
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.0 (4.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 98
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders According to the Modified Teacher's Drooling Scale (mTDS)
Description: The primary efficacy variable was patient's response status using the change from baseline to Week 24 evaluations of the mTDS assessment. Each patient was classified as a responder or non-responder according to the change in their mean mTDS rating from baseline to Week 24. Responders were patients who had at least a 3-point decrease in mTDS rating from baseline
Time Frame: 6 months
Population: The analysis was done by intention to treat method. For purposes of statistical estimation, patients who dropped out due to lack of efficacy had their worst observation carried forward. Patients who dropped out for reasons other than lack of efficacy had their last observation carried forward
Measure: Number; unit: Participants
Arm/Group | Patients With Chronic Drooling
Number analyzed (Participants) | 137
Participants
  Responders | 68
  Non-Responders | 62
  Missing | 7

2. Secondary Outcome: Parent/Caregiver's Assessment of the Extent of Drooling Using Visual Analog Scale (VAS)
Description: Parents/caregivers were to complete a 10 cm "Parent/Caregiver's Assessment of Extent of Drooling for the Day" VAS assessment (0 = normal; 10 = extremely wet) to provide an overall assessment of the extent of drooling for that day.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: VAS score
Arm/Group | Patients With Chronic Drooling
Number analyzed (Participants) | 137
VAS score | 6.56 (2.34)

3. Secondary Outcome: Parent/Caregiver's Assessment of the Extent of Drooling Using VAS
Description: as for outcome 2
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: VAS score
Arm/Group | Patients With Chronic Drooling
Number analyzed (Participants) | 137
VAS score | 3.21 (2.20)

4. Secondary Outcome: Parent/Caregiver's Global Assessment of Treatment
Description: The parent/caregiver performed an overall evaluation of glycopyrrolate liquid for the treatment of drooling, benefits, and side effects over the duration of the study. The parent/caregiver selected one of the following choices to assess if 'This is a worthwhile treatment': 1 = strongly agree, 2 = agree, 3 = neutral, 4 = disagree, 5 = strongly disagree. A dichotomous global assessment was also performed and summarized with the categories 'responder' (strongly agree and agree responses aggregated) and 'non-responder'(neutral, disagree, and strongly disagree responses aggregated)
Time Frame: Week 24
Population: The analysis for parent/caregiver's Global Assessment was done by intention to treat method
Measure: Number; unit: Participants
Arm/Group | Patients With Chronic Drooling
Number analyzed (Participants) | 137
Participants
  Responders | 101
  Non-Responders | 20
  Missing | 16

5. Secondary Outcome: Investigator's Global Assessment of Treatment
Description: The investigator performed an overall evaluation of glycopyrrolate liquid for the treatment of drooling, benefits, and side effects over the duration of the study. The investigator selected one of the following choices to assess if 'This is a worthwhile treatment': 1 = strongly agree, 2 = agree, 3 = neutral, 4 = disagree, 5 = strongly disagree. A dichotomous global assessment was also performed and summarized with the categories 'responder' (strongly agree and agree responses aggregated) and 'non-responder' (neutral, disagree, and strongly disagree responses aggregated)
Time Frame: Week 24
Population: The analysis for investigator's Global Assessment was done by intention to treat method
Measure: Number; unit: Participants
Arm/Group | Patients With Chronic Drooling
Number analyzed (Participants) | 137
Participants
  Responders | 109
  Non-Responders | 18
  Missing | 10

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With Chronic Drooling
Serious Adverse Events (participants affected / at risk) | 14/137
Other Adverse Events (participants affected / at risk) | 122/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Chronic Drooling (N=137)
Nystagmus (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Esophageal candidiasis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) — The serious adverse event of cellulitis was not related to the study drug
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Chronic Drooling (N=137)
Constipation (Gastrointestinal disorders) | 28
Diarrhea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 24
Dry mouth (Gastrointestinal disorders) | 15
Lip dry (Gastrointestinal disorders) | 5
Otitis media (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 11
Influenza (Infections and infestations) | 7
Pharyngitis streptococcal (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 6
Gastroenteritis viral (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 6
Convulsion (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 7
Headache (Nervous system disorders) | 6
Pyrexia (General disorders) | 20
Irritability (General disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 11
Feeding tube complication (Injury, poisoning and procedural complications) | 5
Procedural pain (Injury, poisoning and procedural complications) | 5
Flushing (Vascular disorders) | 15
Restlessness (Psychiatric disorders) | 5
Urine output decreased (Investigations) | 5
Dysuria (Renal and urinary disorders) | 9

LIMITATIONS AND CAVEATS:
There were no limitations of the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.